CLINICAL TRIAL: NCT04640467
Title: Prediction of Late Fetal Growth Restriction in Uncomplicated Pregnancies Using Cerebroplacental Ratio: a Prospective Cohort Study
Brief Title: Prediction of Late Fetal Growth Restriction Using Cerebroplacental Ratio
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Sobhy Shawky, Resident of Obstetrics & Gynecology, Assiut University
Other Study IDs: CPR in late growth restriction
Record Dates: First submitted 2020-09-19; First posted 2020-11-23 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Fetal Growth Retardation; Stillbirth; Neonatal Respiratory Failure; Neonatal Death
Keywords: Cerebroplacental ratio; Fetal growth restriction; Term pregnancy; Doppler ultrasound
MeSH Terms: conditions — Fetal Growth Retardation; Stillbirth; Perinatal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Women with uncomplicated singleton pregnancy who are planning a vaginal delivery, gestational age from 36 ± 0/7 weeks until onset of active labor (cervical dilatation ≤ 4cm) and cephalic presentation
  Interventions: Diagnostic Test: Biophsical profile; Diagnostic Test: Cerebroplacental ratio

INTERVENTIONS:
Diagnostic Test: Biophsical profile — There are five components measured during the biophysical examination. A score of 2 points is given for each component that meets criteria. The test is continued until all criteria are met or 30 minutes have elapsed. The points are then added for a possible maximum score of 10. A total score of 10 out of 10 or 8 out of 10 with normal fluid is considered normal. A score of 6 is considered equivocal, and a score of 4 or less is abnormal.
  Other Names: BPP
Diagnostic Test: Cerebroplacental ratio — CPR is the ratio of the Middle Cerebral Artery Pulsatility Index (MCA PI) to the Umbilical Artery Pulsatility Index (UA PI). The pulsatility indices will be measured from an automated trace of at least three consecutive waveforms of the relevant vessel in the absence of fetal breathing movements or uterine contractions. The angle of insonation will be as close to zero degrees as possible. The UA PI will be recorded from a free-floating section of cord, and the MCA PI will be obtained from the proximal third of the vessel (10, 14).
  Other Names: CPR

SUMMARY:
To investigate the screening performance of CPR and biophysical profile score for the prediction of composite of adverse neonatal morbidity and mortality and operative delivery (CS or instrumental) for intrapartum fetal distress in low-risk pregnancies

DETAILED DESCRIPTION:
Fetal growth is a dynamic process and its assessment requires multiple observations over time. In most women, placental function is sufficient to allow appropriate fetal growth throughout pregnancy, however in some, it may be not near term or during labor leading to intrapartum compromise Small for gestational age (SGA) is estimated fetal weight (EFW) or abdominal circumference (AC) below the 10th percentile of given reference ranges Fetal growth restriction (FGR) is fetus that has not achieved its growth potential. There are early-onset (< 32 weeks) and late-onset (≥ 32 weeks) types. Late FGR is defined as

- AC/EFW < 3rd centile Or at least two out of three of:

1. AC/EFW < 10th centile
2. AC/EFW crossing centiles >2 quartiles
3. Cerebroplacental ratio (CPR) <5th centile or Umbilical artery Pusitility Index(UAPI )>95th centile FGR fetuses will not necessarily be SGA at delivery and vice versa. In fact, most SGA are likely to be 'constitutionally' small CPR is the ratio of the Middle cerebral artery Pulsatility Index (MCAPI) to (UAPI). The CPR gradually rises until around the 34th week and subsequently slowly declines until term. Its use has been echoed recently because of association of an abnormal ratio with fetal distress in labor requiring emergency cesarean section , a lower cord pH, admission to the intensive care unit and poor neurological outcomes The biophysical profile (BPP) abnormalities that characterize late FGR include alteration of fetal breathing, oligohydramnios and loss of fetal heart rate reactivity on conventional cardiotocography ( CTG). It seems that BPP becomes abnormal only shortly before stillbirth .

ELIGIBILITY:
Inclusion Criteria:

* •Women with uncomplicated singleton pregnancy who are planning a vaginal delivery

  * Gestational age from 36 ± 0/7 weeks until onset of active labor (cervical dilatation ≤ 4cm)
  * Cephalic presentation

Exclusion Criteria:

* •Multiple pregnancy

  * known SGA fetus.
  * Medical disorders with pregnancy: diabetes mellitus, hypertension, pre-eclampsia
  * Known fetal anomaly or aneuploidy or stillbirth.
  * Any contraindication of vaginal delivery eg. placenta previa.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Women with uncomplicated singleton pregnancy who are planning a vaginal delivery.
  Gestational age from 36 ± 0/7 weeks until onset of active labor (cervical dilatation ≤ 4cm) with cephalic presentation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
A composite of adverse neonatal outcomes | Up to 48 hours After delivery
  Apgar score ≤7 at 5 min or resuscitation with intubation, chest compressions or medication, admission to NICU ≥ 48 hours or hypoxic ischemic encephalopathy or cerebral palsy or stillbirth or neonatal death within 28 days

SECONDARY OUTCOMES:
Operative delivery (instrumental and caesarean section) for intrapartum fetal compromise (IFC) | At time of delivery
  The diagnosis of IFC will be made by the treating obstetrician based on abnormal fetal heart rate patterns (classified according to National Institute for Health and Clinical excellence [NICE] guidelines ) (15) or presence of meconium stained liquor.
Demographic characteristics of the cohort | Gestational age from 36 ± 0/7 weeks until onset of active labor (cervical dilatation ≤ 4cm)
  Demographic characteristics of the cohort
Estimated fetal weight | At Ultrasound examination at Gestational age from 36 ± 0/7 weeks until onset of active labor (cervical dilatation ≤ 4cm)
  An ultrasonographic measurement using Hadlock formula (13)
Birth weight | Immediatly after delivery
  Birth weight in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Sobhy, MBBCH, Principal Investigator — Assiut University; Ahmed Aboelhasan, MD, Principal Investigator — Assiut University; Moustafa Gadalla, MD, Principal Investigator — Assiut University
Locations (1):
- Women's Health Hospital, Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Sherrell H, Clifton V, Kumar S. Predicting intrapartum fetal compromise at term using the cerebroplacental ratio and placental growth factor levels (PROMISE) study: randomised controlled trial protocol. BMJ Open. 2018 Aug 13;8(8):e022567. doi: 10.1136/bmjopen-2018-022567. PMID 30104317
- [Background] Lees CC, Stampalija T, Baschat A, da Silva Costa F, Ferrazzi E, Figueras F, Hecher K, Kingdom J, Poon LC, Salomon LJ, Unterscheider J. ISUOG Practice Guidelines: diagnosis and management of small-for-gestational-age fetus and fetal growth restriction. Ultrasound Obstet Gynecol. 2020 Aug;56(2):298-312. doi: 10.1002/uog.22134. No abstract available. PMID 32738107
- [Background] Gordijn SJ, Beune IM, Thilaganathan B, Papageorghiou A, Baschat AA, Baker PN, Silver RM, Wynia K, Ganzevoort W. Consensus definition of fetal growth restriction: a Delphi procedure. Ultrasound Obstet Gynecol. 2016 Sep;48(3):333-9. doi: 10.1002/uog.15884. PMID 26909664
- [Background] Monier I, Blondel B, Ego A, Kaminiski M, Goffinet F, Zeitlin J. Poor effectiveness of antenatal detection of fetal growth restriction and consequences for obstetric management and neonatal outcomes: a French national study. BJOG. 2015 Mar;122(4):518-27. doi: 10.1111/1471-0528.13148. Epub 2014 Oct 27. PMID 25346493
- [Background] Ebbing C, Rasmussen S, Kiserud T. Middle cerebral artery blood flow velocities and pulsatility index and the cerebroplacental pulsatility ratio: longitudinal reference ranges and terms for serial measurements. Ultrasound Obstet Gynecol. 2007 Sep;30(3):287-96. doi: 10.1002/uog.4088. PMID 17721916
- [Background] Cruz-Martinez R, Figueras F, Hernandez-Andrade E, Oros D, Gratacos E. Fetal brain Doppler to predict cesarean delivery for nonreassuring fetal status in term small-for-gestational-age fetuses. Obstet Gynecol. 2011 Mar;117(3):618-626. doi: 10.1097/AOG.0b013e31820b0884. PMID 21343765
- [Background] Stampalija T, Thornton J, Marlow N, Napolitano R, Bhide A, Pickles T, Bilardo CM, Gordijn SJ, Gyselaers W, Valensise H, Hecher K, Sande RK, Lindgren P, Bergman E, Arabin B, Breeze AC, Wee L, Ganzevoort W, Richter J, Berger A, Brodszki J, Derks J, Mecacci F, Maruotti GM, Myklestad K, Lobmaier SM, Prefumo F, Klaritsch P, Calda P, Ebbing C, Frusca T, Raio L, Visser GHA, Krofta L, Cetin I, Ferrazzi E, Cesari E, Wolf H, Lees CC; TRUFFLE-2 Group. Fetal cerebral Doppler changes and outcome in late preterm fetal growth restriction: prospective cohort study. Ultrasound Obstet Gynecol. 2020 Aug;56(2):173-181. doi: 10.1002/uog.22125. PMID 32557921
- [Background] Crimmins S, Desai A, Block-Abraham D, Berg C, Gembruch U, Baschat AA. A comparison of Doppler and biophysical findings between liveborn and stillborn growth-restricted fetuses. Am J Obstet Gynecol. 2014 Dec;211(6):669.e1-10. doi: 10.1016/j.ajog.2014.06.022. Epub 2014 Jun 12. PMID 24931475
- [Background] Khalil AA, Morales-Rosello J, Morlando M, Hannan H, Bhide A, Papageorghiou A, Thilaganathan B. Is fetal cerebroplacental ratio an independent predictor of intrapartum fetal compromise and neonatal unit admission? Am J Obstet Gynecol. 2015 Jul;213(1):54.e1-54.e10. doi: 10.1016/j.ajog.2014.10.024. Epub 2014 Oct 18. PMID 25446667
- [Background] Bligh LN, Alsolai AA, Greer RM, Kumar S. Prelabor screening for intrapartum fetal compromise in low-risk pregnancies at term: cerebroplacental ratio and placental growth factor. Ultrasound Obstet Gynecol. 2018 Dec;52(6):750-756. doi: 10.1002/uog.18981. PMID 29227010
- [Background] Practice bulletin no. 145: antepartum fetal surveillance. Obstet Gynecol. 2014 Jul;124(1):182-192. doi: 10.1097/01.AOG.0000451759.90082.7b. No abstract available. PMID 24945455
- [Background] Manning FA. The fetal biophysical profile score: current status. Obstet Gynecol Clin North Am. 1990 Mar;17(1):147-62. PMID 2192316
- [Background] Hadlock FP, Harrist RB, Martinez-Poyer J. In utero analysis of fetal growth: a sonographic weight standard. Radiology. 1991 Oct;181(1):129-33. doi: 10.1148/radiology.181.1.1887021.
- [Background] Baschat AA, Gembruch U. The cerebroplacental Doppler ratio revisited. Ultrasound Obstet Gynecol. 2003 Feb;21(2):124-7. doi: 10.1002/uog.20. PMID 12601831
- [Background] Kenyon S, Ullman R, Mori R, Whittle M. Care of healthy women and their babies during childbirth: summary of NICE guidance. BMJ. 2007 Sep 29;335(7621):667-8. doi: 10.1136/bmj.39322.703380.AD. No abstract available. PMID 17901518